CLINICAL TRIAL: NCT03722368
Title: An Evaluation of a Tiered Approach to Increase Well-Being in Healthcare and Social Service Providers in a Post-Disaster Context
Brief Title: Health and Wellness in Healthcare Providers Post-disaster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Americares (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Colorado State University (Other)
Responsible Party: Principal Investigator, Tara Powell, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 18699
Record Dates: First submitted 2018-10-16; First posted 2018-10-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Intervention 1: Resilience and Coping for Healthcare Group; Intervention 2: Resilience and Coping for Healthcare Plus Additional Services; Waitlist Control Group
MeSH Terms: interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RCHC (Experimental): Participation in the Resilience and Coping of the Healthcare Community Intervention.
  Interventions: Behavioral: RCHC
- RCHC+ (Experimental): Participation in the Resilience and Coping of the Healthcare Community Intervention, support groups and one on one counseling.
  Interventions: Behavioral: RCHC+
- Waitlist Control (Other): This group will receive treatment as usual and will be offered services once the study is complete.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: RCHC — The RCHC group will receive a three hour psychoeducational intervention on common stress responses among healthcare providers and coping skills. They will also receive a booster session one month later which will reinforce these skills.
  Arms: RCHC
Behavioral: RCHC+ — The RCHC group will receive a three hour psychoeducational intervention on common stress responses among healthcare providers and coping skills. They will also receive a booster session one month later which will reinforce these skills. This intervention group will also receive on-going support groups and one on one counseling as needed.
  Other Names: Resilience and Coping for the Healthcare Community Plus additional Services
  Arms: RCHC+
Other: Waitlist control — This group will served as the control group and will receive treatment as usual until the end of the study. At the end of the study they will have the opportunity to take part in the RCHC or RCHC+
  Arms: Waitlist Control

SUMMARY:
The purpose of this evaluation is to understand the impact of mental health and psychosocial support (MHPS) programming that AmeriCares (a non-profit disaster response organization) is currently providing to healthcare and social service providers in Southeast Texas and Puerto Rico. The MHPS services are designed to provide skills to reduce stress, improve coping and reduce symptoms of burnout (compassion fatigue).

DETAILED DESCRIPTION:
Health care and social service providers from disaster-affected communities are at heightened risk for emotional distress symptoms immediately after the event and over the longer-term recovery period. They provide care to others both physically and emotionally, while at the same time are often in the process of recovery and rebuilding their own lives. Health care providers, particularly those who work in safety net health centers, often serve high-need communities where incomes are lower, health issues are elevated, and health care is scarce.

Given the high risk for emotional distress symptoms for healthcare workers after a disaster, it is critical to offer services to help ease the stress during the hurricane recovery. This evaluation will examine the impact of Americares mental health and psychosocial (MHPS) programming on care providers in the short- and longterm recovery. The purpose of this evaluation is to understand the impact of mental health and psychosocial support (MHPS) programming that AmeriCares (a non-profit disaster response organization) is currently providing to healthcare and social service providers in Southeast Texas and Puerto Rico. The MHPS services are designed to provide skills to reduce stress, improve coping and reduce symptoms of burnout (compassion fatigue).

The study included naturalistic groups that will receive services from Americares based on the agencies needs.

They will include:

1. A waitlisted control group who will receive services within 3-months after the study begins
2. A group who will receive one specific workshop, known as RCHC (Resilience and Coping for the Healthcare Community)
3. A group who will receive RCHC plus additional services (RCHC+)

The 3-hour RCHC intervention draws from existing literature and theory on effective psychosocial interventions and integrates the following components:

* An open interactive learning environment
* A safe environment for open communication
* Education and strategies to support highly stressed and/or traumatized patients.
* Psycho-education about stress and coping
* Planning for coping strategies
* Identification and referral to mental health resources The additional services will include wellness groups and psychoeducational training. The wellness groups include a variety of topics, designed to promote healthy living and empowerment. Each one-hour group will be facilitated by Americares staff and tailored to particular needs of the group. Topics may include but not limited to: Grief and loss, Stress management, Workplace wellness, Navigating support systems. The psychoeducational trainings provide healthcare workers with educational resources to support their patients in the aftermath of Harvey and recognize and respond to stress reactions. Training topics include: Psychological First Aid for Adults, Psychological First Aid for Children, The Brain, the Body and Trauma, Coping with Difficult Workplace Situations.

ELIGIBILITY:
Inclusion criteria:

Healthcare workers will be eligible for the study if they are:

1. over 18 years of age at the time of admission into the study;
2. speak and read English or Spanish;
3. have been identified as having experienced Hurricane Harvey or Maria or providing care to people living in areas affected by the storms;
4. are employed by a participating Community Health Center or partnering agency;
5. participate in AmeriCares MHPS programs.

Exclusion criteria: Healthcare workers will be excluded if they:

1. do not meet the inclusion criteria, or
2. do not give consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
ProQol--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  The ProQOL 5 is a 30-item scale for measuring professional quality of life among people who work in the helping professions (Stamm, 2010). The tool measures the positive aspect of compassion satisfaction (the pleasure you derive from being able to do your work well), and the negative aspect of compassion fatigue, which is composed of two parts: burnout (exhaustion, frustration and anger) and secondary trauma (work-related secondary exposure to people who have experienced traumatic events).

SECONDARY OUTCOMES:
Social Provisions Scale--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  Subscales of the Social Provisions Scale (SPS) (Cutrona & Russel, 1987) (8 items): Reliable Alliance (4), Guidance (4) For the purposes of our study, the instructions leading into the SPS were changed to restrict participants to thinking about co-workers. The measure asks respondents to rate the degree to which their social relationships are currently supplying each of the provisions. Each provision is assessed by four items, two that describe the presence and two that describe the absence of the provision. Respondents indicate on 4-point scales (ranging fromcompletely true to not at all true ) the extent to which each statement describes their current social relationships. For scoring purposes, the negative items are reversed and summed together with the positive items to form a score for each social provision. Reliability for the total support score in a previous study was .92, with reliabilities of the 4-item subscales ranging from .76 to .84 (Cutrona, Russell, & Rose, 1986).
Brief Resilience Scale--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  The brief resilience scale (BRS) was created to assess the ability to bounce back or recover from stress. The BRS has been tested and is reliable as a unitary construct. It is predictably related to personal characteristics, social relations, coping, and health in all samples. It was negatively related to anxiety, depression, negative affect, and physical symptoms when other resilience measures and optimism, social support.
Perceived Stress Scale (PSS) (10)--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  The PSS is a widely used measure of the degree to which situations in one's life are appraised as stressful (Cohen, Kessler, & Underwood Gordon, 1994) .
Impact of Events Scale-Revised--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  Six item screen derived from the PTSD Checklist-Civilian Version to help primary care settings screen for persons with possible PTSD symptoms. The six items evaluate reexperiencing, avoidance, and hyperarousal which are highly correlated with the PCL-C. The full checklist was studied and utilized to screen for PTSD in countries such as China , Armenia, and Nepal.
Brief Cope--Assessing change over time | Baseline, 6 weeks, 12 weeks, 18 weeks
  The Brief COPE measures 14 identified coping responses: Self-distraction, Active coping, Denial, Substance use, use of instrumental support, use of emotional support, behavioral disengagement, venting, positive reframing, acceptance, planning, humor, religion, and Self-blame. It represents a way to rapidly measure coping responses because it is a short 28-item self-report questionnaire with two items for each of the measured coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Powell, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- Americares, Houston, Texas, United States
- Americares Puerto Rico, San Juan, Puerto Rico